CLINICAL TRIAL: NCT03880019
Title: A Phase II Study of the PARP Inhibitor Olaparib in Combination With the DNA Damaging Agent Temozolomide for the Treatment of Advanced Uterine Leiomyosarcoma
Brief Title: A Phase II Clinical Trial Evaluating the Combination of Olaparib and Temozolomide for the Treatment of Advanced Uterine Leiomyosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01500; NCI-2019-01500 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); #AAAS4040; WUSM HRPO# 201910106; 10250 (Other: Yale University Cancer Center LAO); 10250 (Other: CTEP); UM1CA186686 (NIH)
Record Dates: First submitted 2019-03-18; First posted 2019-03-19 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Stage III Uterine Corpus Leiomyosarcoma AJCC v8; Stage IV Uterine Corpus Leiomyosarcoma AJCC v8; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — Biopsy, Needle; Biopsy, Large-Core Needle; Magnetic Resonance Spectroscopy; olaparib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib, temozolomide) (Experimental): Patients receive olaparib PO BID and temozolomide PO QD on days 1-7 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI throughout the trial and undergo tumor biopsy at screening and on study.
  Interventions: Procedure: Computed Tomography; Procedure: Core Biopsy; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Drug: Temozolomide

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Core Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY, CORE; CNB; Core Needle; Core Needle Biopsy; Needle Biopsy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial studies olaparib and temozolomide in treating patients with uterine leiomyosarcoma (LMS) that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced), that has spread from where it first started to other places in the body (metastatic) or cannot be removed by surgery (unresectable). PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving olaparib and temozolomide may work better than giving either drug alone in treating patients with LMS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether combination treatment with temozolomide (TMZ) + olaparib shows preliminary evidence of clinical activity among patients with advanced uterine leiomyosarcoma (LMS) as measured by the confirmed objective response rate (ORR).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile associated with the combination treatment. II. To evaluate the progression free survival (PFS) associated with the combination treatment.

III. To evaluate what proportion of uterine LMS tumors exhibit homologous recombination (HR) deficiency as measured by (1) genomic alterations in HR components at baseline and (2) deoxyribonucleic acid (DNA) repair protein RAD51 homolog (RAD51) foci formation at baseline and while on study treatment.

IV. To evaluate the feasibility of these assays in human tissue, and to preliminarily evaluate for any association between presence of HR deficiency as measured by each assay and increased clinical benefit from the study treatment.

EXPLORATORY OBJECTIVES:

I. To evaluate what proportion of uterine LMS tumors exhibit HR deficiency as measured by Schlafen family member number 11(SLFN11) protein expression at baseline.

II. To evaluate the feasibility of this assay in human tissue, and to preliminarily evaluate for any association between presence of HR deficiency as measured by this assay and increased clinical benefit from the study treatment.

III. To evaluate MGMT protein expression in uterine LMS tumors, and to preliminarily evaluate for any association between MGMT expression and increased clinical benefit from the study treatment.

IV. To perform an optional third tissue biopsy in patients who initially benefit from study treatment but later show early evidence of disease progression to evaluate for changes in the status of the RAD51 foci, MGMT, and SLFN11 assays at that time.

OUTLINE:

Patients receive olaparib orally (PO) twice per day (BID) and temozolomide PO once daily (QD) on days 1-7 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial and undergo tumor biopsy at screening and on study.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then every 6 months until death or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented LMS of uterine origin. Pathology review and confirmation of diagnosis will occur at the site enrolling the patient on this study.
* Patients must have locally advanced and unresectable or metastatic disease.
* Patients must have disease which is measurable at study entry according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. Additionally, patients must have a site of disease deemed accessible for biopsy at no or minimal risk to the patient (including through the use of image-guidance). If there are questions regarding the feasibility of biopsy, the case should be reviewed with interventional radiology or the appropriate department at the study site prior to registration.
* Patients must have had prior progression on, or intolerance to, at least one line of systemic therapy for advanced LMS. Adjuvant therapy administered after curative resection will not qualify as prior treatment. There is no upper limit on the number of prior therapies received.
* Patients must be >= 18 years of age. Uterine LMS affects older adults and is rarely encountered in children and adolescents.
* Patients must demonstrate an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of =< 2 (Karnofsky >= 50%).
* Absolute neutrophil count >= 1,500/mcL (measured within 14 days prior to administration of study treatment).
* Hemoglobin >= 9 g/dL (without transfusion of packed red blood cells within the past 28 days) (measured within 14 days prior to administration of study treatment).
* Platelets >= 100,000/mcL (measured within 14 days prior to administration of study treatment).
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (measured within 14 days prior to administration of study treatment).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (measured within 14 days prior to administration of study treatment).
* Glomerular filtration rate (GFR) >= 51 mL/min, based on a 24-hour urine test for creatinine clearance or estimated using the Cockcroft-Gault equation (measured within 14 days prior to administration of study treatment).
* If patients have evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of hepatitis B surface antigen [HBsAg]) are eligible.
* If patients have a history of hepatitis C virus (HCV) infection, they must be treated with undetectable HCV viral load (polymerase chain reaction is negative for HCV ribonucleic acid [RNA]).
* Patients must be postmenopausal or have evidence of non-childbearing status, OR, for women of childbearing potential, must have a negative urine or serum pregnancy test within 28 days of study treatment and confirmed again on day 1 prior to study treatment.

  * Postmenopausal is defined as:

    * Amenorrheic for >= 1 year following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50
    * Radiation-induced oophorectomy with last menses > 1 year ago
    * Chemotherapy-induced menopause with > 1 year interval since last menses
    * Surgical sterilization (bilateral oophorectomy or hysterectomy).
* Patients and their partners, if sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for 3 months after the last dose of study drug(s) to prevent pregnancy in the study patient or partner.
* Patients must be able to swallow orally administered medication.
* Patients must have a life expectancy >= 16 weeks.
* Patients must be able to understand and be willing to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) will be eligible if they have a close caregiver or legally authorized representative (LAR) available to assist them.
* Patients must be willing and able to comply with the protocol for the duration of the study, including undergoing treatment and attending scheduled visits and examinations.
* Patients with human immunodeficiency virus (HIV) infection may be enrolled on this study provided: (a) they are on a stable regimen of highly active anti-retroviral therapy (HAART) with no medications otherwise prohibited by this protocol (e.g. drug-drug interactions) and (b) require no concurrent antibiotics or antifungals for the prevention of opportunistic infections and (c) have a CD4 count above 250 cell/mcL and an undetectable viral load on standard polymerase chain reaction (PCR)-based tests within 1 month of initiation of study treatment. Other patients with clinically significant immunosuppression, e.g. organ transplant patients, are not eligible. If clarification is needed, this may be discussed with the medical monitor.
* Patients must be able to have temozolomide provided as a standard of care medication.

Exclusion Criteria:

* Patients must not have had any previous treatment with any poly(adenosine diphosphate[ADP]-ribose) polymerase (PARP) inhibitors, including olaparib, or prior treatment with dacarbazine and/or temozolomide.
* Patients must have recovered from adverse events due to prior anti-cancer therapy (i.e., may not have residual toxicities > grade 1 or above baseline), excluding alopecia. Patients who have endocrinopathies associated with prior immunotherapy treatment but which are controlled with replacement therapy are eligible.
* Prior to initiating study treatment, at least 28 days must have elapsed from the last dose of systemic anti-cancer treatment (cytotoxic, biologic or immunotherapeutic) or radiation therapy (except for palliative radiation, in which case a 14-day washout applies).
* Patients must not have had major surgery within 2 weeks of starting study treatment and must have recovered from any effects of any major surgery that occurred > 2 weeks before starting study treatment.
* Patients must not be receiving any other investigational agent.
* Patients must not have been diagnosed with another malignancy unless curatively treated with no evidence of disease for >= 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), or any other malignant condition considered indolent and unlikely to require active therapy.
* Patients must not have myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or bone marrow biopsy findings consistent with MDS and/or AML.
* Patients must not have active central nervous system (CNS) or leptomeningeal disease at the time of enrollment. Patients with a history of such disease previously treated with curative intent (such as with surgery or radiation) that have not progressed on subsequent imaging, have been clinically asymptomatic, and have not received systemic corticosteroids for at least 28 days, are eligible.
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib or TMZ or any of the excipients of any study product.
* Patients must refrain from concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period for strong or moderate CYP3A inhibitors prior to starting olaparib is 2 weeks. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patients must refrain from concomitant use of known strong CYP3A inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil). The required washout period for strong or moderate CYP3A inducers prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patients must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan, or psychiatric illness that would limit compliance with study requirements.
* Pregnant women are excluded from this study because olaparib is a PARP inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib, breastfeeding should be discontinued if the mother is treated with olaparib. These potential risks may also apply to other agents used in this study.
* Patients must not have gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients must not have had involvement in the planning and/or conduct of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2026-11-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mia C Weiss, Principal Investigator — Yale University Cancer Center LAO
Locations (15):
- United States (15):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Ingham M, Allred JB, Chen L, Das B, Kochupurakkal B, Gano K, George S, Attia S, Burgess MA, Seetharam M, Boikos SA, Bui N, Chen JL, Close JL, Cote GM, Thaker PH, Ivy SP, Bose S, D'Andrea A, Marino-Enriquez A, Shapiro GI, Schwartz GK. Phase II Study of Olaparib and Temozolomide for Advanced Uterine Leiomyosarcoma (NCI Protocol 10250). J Clin Oncol. 2023 Sep 1;41(25):4154-4163. doi: 10.1200/JCO.23.00402. Epub 2023 Jul 19. PMID 37467452
- [Derived] Vyse S, Thway K, Huang PH, Jones RL. Next-generation sequencing for the management of sarcomas with no known driver mutations. Curr Opin Oncol. 2021 Jul 1;33(4):315-322. doi: 10.1097/CCO.0000000000000741. PMID 33927108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One enrolled patient did not begin treatment.
Groups:
- Treatment (Olaparib, Temozolomide): Patients receive olaparib PO BID and temozolomide PO QD on days 1-7. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI once every 2 cycles. For patients who continue beyond 12 cycles, MRI or CT imaging may be changed to once every 4 cycles. Patients undergo tumor biopsy cycle 2 days 3-5.
  >
  > Computed Tomography: Undergo CT
  >
  > Core Biopsy: Undergo tumor biopsy
  >
  > Magnetic Resonance Imaging: Undergo MRI
  >
  > Olaparib: Given orally (PO)
  >
  > Temozolomide: Given PO
Period: Overall Study
Arm/Group | Treatment (Olaparib, Temozolomide)
Started | 23
Completed | 22
Not Completed | 1
Not completed — Competing disease | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Olaparib, Temozolomide): Patients receive olaparib PO BID and temozolomide PO QD on days 1-7. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI once every 2 cycles. For patients who continue beyond 12 cycles, MRI or CT imaging may be changed to once every 4 cycles. Patients undergo tumor biopsy cycle 2 days 3-5.>
  > Computed Tomography: Undergo CT>
  > Core Biopsy: Undergo tumor biopsy>
  > Magnetic Resonance Imaging: Undergo MRI>
  > Olaparib: Given orally (PO)>
  > Temozolomide: Given PO
Arm/Group | Treatment (Olaparib, Temozolomide)
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 55 [39 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Stage at Study Entry [Count of Participants; unit: Participants]
  Locally advanced/unresectable | 3
  Metastatic | 17
  Unknown | 2
Prior Lines of Treatment [Count of Participants; unit: Participants]
  1-2 | 9
  3 or more | 13
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 7
    1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) (Complete Response + Partial Response)
Description: Will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria assessed by MRI: Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm); Partial Response (PR), at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. A response rate of 10% is considered inactive and unworthy of further study. A response rate of 35% would be promising for further study among patients with advanced uterine leiomyosarcoma (LMS) treated with at least one prior systemic regimen. A response rate of 35% for the temozolomide (TMZ) + poly(adenosine diphosphate[ADP]-ribose) polymerase inhibitor (PARPi) combination would also be suggestive of superior efficacy over TMZ monotherapy in sarcoma. Will be reported with a 95% confidence interval.
Time Frame: Within first 6 months of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib, Temozolomide)
Number analyzed (Participants) | 22
Participants | 5

2. Secondary Outcome: Number of Patients Experiencing Adverse Events
Description: Recorded at each clinical visit and will be categorized according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Number of patients experiencing a grade 3 or greater adverse event will be reported.
Time Frame: Up to 2 years after study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Olaparib, Temozolomide)
Number analyzed (Participants) | 22
Participants | 20

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The Kaplan-Meier method will be used to evaluate time to event endpoints. Median PFS will be reported with a 95% confidence interval.
Time Frame: Time from first treatment with the study drug to the earliest of either disease progression or death from any cause, assessed up to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Uterine LMS Tumors Exhibit Homologous Recombination (HR) Deficiency
Description: Will be measured by genomic alterations in HR components at baseline and deoxyribonucleic acid (DNA) repair protein RAD51 homolog (RAD51) foci formation. The two integrated assays are genomics for alterations in HR genes and RAD51 foci formation. Both of these assays report binary results. The rate of response will be compared between binary variables using the Fisher's exact test. The log-rank test will be used to compare PFS between binary variables. Additional results from whole exome sequencing and ribonucleic acid sequencing (RNAseq) analysis on study samples will be reported in a descriptive fashion.
Time Frame: Up to 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Schlafen Family Member Number 11(SLFN11) Protein Expression
Description: Will be assessed by immunohistochemistry (ICH). Macro ribonucleic acid (mRNA) expression may also be performed. Expression are reported as a continuous variable. Logistic regression will be used to estimate the odds of response for every unit increase in protein expression. Cox-regression will be used to evaluate the association between PFS and protein expression. Graphical displays such as box plots and Kaplan-Meier plots will be used to visualize the data. Evaluate for any association between presence of HR deficiency and increased clinical benefit from study treatment.
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of MGMT Protein Expression in Uterine LMS Tumors
Description: Will be assessed by ICH. mRNA expression may also be performed. Expression are reported as a continuous variable. Logistic regression will be used to estimate the odds of response for every unit increase in protein expression. Cox-regression will be used to evaluate the association between PFS and protein expression. Graphical displays such as box plots and Kaplan-Meier plots will be used to visualize the data. Evaluate for any association between MGMT expression and increased clinical benefit from the study treatment.
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 34 months
Arm/Group | Treatment (Olaparib, Temozolomide)
All-Cause Mortality (participants affected / at risk) | 8/22
Serious Adverse Events (participants affected / at risk) | 19/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Olaparib, Temozolomide) (N=22)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 16 (28)
Platelet count decreased (Investigations) | 7 (12)
Sinus tachycardia (Cardiac disorders) | 1 (1)
White blood cell decreased (Investigations) | 5 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Olaparib, Temozolomide) (N=22)
Abdominal pain (Gastrointestinal disorders) | 6 (26)
Abdominal tenderness near umbilicus (Gastrointestinal disorders) | 1 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (8)
Alanine aminotransferase increased (Investigations) | 2 (7)
Alkaline phosphatase increased (Investigations) | 5 (24)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (21)
Anal fissure (Gastrointestinal disorders) | 1 (18)
Anemia (Blood and lymphatic system disorders) | 16 (188)
Anorexia (Metabolism and nutrition disorders) | 6 (22)
Anxiety (Psychiatric disorders) | 1 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (36)
Aspartate aminotransferase increased (Investigations) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (45)
Blepharospasm (left eye) (Eye disorders) | 1 (4)
Blood bicarbonate decreased (Investigations) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 3 (16)
Blurred vision (Eye disorders) | 1 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (19)
Breast pain (Reproductive system and breast disorders) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Cold flashes (General disorders) | 1 (2)
Cold flashes, intermittent (General disorders) | 1 (11)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (61)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Creatinine increased (Investigations) | 4 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 9 (42)
Dizziness (Nervous system disorders) | 5 (31)
Dry mouth (Gastrointestinal disorders) | 2 (32)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (26)
Dysgeusia (Nervous system disorders) | 3 (17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (36)
Dysuria (Renal and urinary disorders) | 1 (3)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 6 (38)
Fatigue (General disorders) | 14 (160)
Fever (General disorders) | 5 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (3)
Flu like symptoms (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Fogginess feeling (General disorders) | 1 (2)
GGT increased (Investigations) | 2 (10)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (48)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (11)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (37)
Hemoglobin decrease (Blood and lymphatic system disorders) | 1 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 2 (2)
Hot flashes (Vascular disorders) | 4 (15)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (55)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (5)
Hypertension (Vascular disorders) | 6 (22)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (15)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 3 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (5)
INR increased (Investigations) | 2 (13)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (49)
L eye irritation (Eye disorders) | 1 (14)
Lymphocyte count decreased (Investigations) | 7 (44)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (16)
Mucositis oral (Gastrointestinal disorders) | 1 (13)
Muscle weakness left-sided (Nervous system disorders) | 1 (9)
Muscle weakness right-sided (Nervous system disorders) | 1 (9)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (16)
Nail infection (Infections and infestations) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (10)
Nausea (Gastrointestinal disorders) | 12 (121)
Neutrophil count decreased (Investigations) | 18 (166)
Oral hemorrhage (Gastrointestinal disorders) | 2 (3)
Oral pain (Gastrointestinal disorders) | 4 (25)
Pain (General disorders) | 4 (27)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (22)
Paresthesia (Nervous system disorders) | 2 (32)
Pelvic pain (Reproductive system and breast disorders) | 1 (9)
Periodontal disease (Gastrointestinal disorders) | 1 (10)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (5)
Platelet count decreased (Investigations) | 19 (185)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (13)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (4)
Sinus bradycardia (Cardiac disorders) | 1 (3)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (18)
Sinus tachycardia (Cardiac disorders) | 3 (9)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stomach Gas (Gastrointestinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (5)
Toothache (Gastrointestinal disorders) | 1 (2)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (3)
Urinary urgency (Renal and urinary disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (22)
Weight gain (Investigations) | 3 (26)
Weight loss (Investigations) | 2 (13)
White blood cell decreased (Investigations) | 17 (190)
nail ridges peeling (Skin and subcutaneous tissue disorders) | 1 (11)
pinching pain near vagina (left side) (General disorders) | 1 (1)
small warty lesion on left labia (Reproductive system and breast disorders) | 1 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03880019/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT03880019/ICF_001.pdf